CLINICAL TRIAL: NCT06546917
Title: The bWell Cognitive Care Platform: A Pilot Feasibility Study in Patients With Depression
Brief Title: bWell-D Pilot Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Simon Fraser University (Other); National Research Council, Canada (Unknown)
Responsible Party: Principal Investigator, Trisha Chakrabarty, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H24-00404
Record Dates: First submitted 2024-07-23; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Depressive Disorder, Major; Cognitive Dysfunction
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are told that either arm is hypothesized to have effects on their cognition and are therefore blinded to whether they are in the 'active' treatment group.
  Assessors for outcomes that are not self-reported or self-administered will also be blinded as to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bWell Cognitive Remediation (Active Comparator): Patients with Major Depressive Disorder who will complete cognitive remediation sessions using bWell twice a week for eight weeks.
  Interventions: Behavioral: bWell Cognitive Remediation
- VR Experience (Sham Comparator): Patients with Major Depressive Disorder who will experience various VR scenes twice a week for eight weeks.
  Interventions: Behavioral: VR Experience

INTERVENTIONS:
Behavioral: bWell Cognitive Remediation — Patients will take part in the bWell cognitive remediation protocol, consisting of 40-minute sessions of bWell, administered 2 times a week for 8 weeks. These sessions consist of tasks that target various cognitive domains and increase in complexity and difficulty as training progresses. The tasks are as follows:
  1. Lab Exercise: participant alternates between two different, increasingly complex 'recipes', targeting executive functioning and divided attention.
  2. Egg Exercise: In an office environment, participants must seek out and maintain their gaze on certain objects in order to collect them in the presence of visual distractors, targeting sustained attention.
  3. Mole Exercise: participants must strike moles with the matching coloured hammer as fast as possible, targeting selective attention.
  4. Theatre Exercise: participants must remember objects presented on stage and recreate the sequence after the curtains close, targeting working memory.
  Arms: bWell Cognitive Remediation
Behavioral: VR Experience — Patients will take part in the viewing of VR scenes which contain no instructed cognitive tasks. This consists of 40-minute sessions of viewing VR scenes, administered 2 times a week for 8 weeks.
  Arms: VR Experience

SUMMARY:
The goal of this clinical trial is to determine the acceptability, feasibility, and validity of the bWell Cognitive Care Platform for Depression (bWell-D), a novel Virtual Reality (VR) cognitive assessment and remediation tool, in depressed populations. The main questions are:

* Do patients with Major Depressive Disorder (MDD) find the bWell-D cognitive assessment battery and protocol feasible, tolerable, and acceptable?
* Do patients with Major Depressive Disorder (MDD) find the 8 week bWell-D remediation protocol feasible, tolerable, and acceptable?

Following initial cognitive assessment, researchers will assess feasibility outcomes in the bWell remediation arm to a VR scenes experience arm to learn more about the feasibility of bWell for cognitive assessment and remediation.

Patients will:

* Complete an initial bWell cognitive assessment session
* Randomized to either receive bWell cognitive remediation or a VR scenes experience twice a week for eight weeks
* Complete cognitive/functional/clinical assessments and EEG at baseline, midpoint and endpoint of the remediation protocol, as well as measures of tolerability, engagement, and enjoyment

DETAILED DESCRIPTION:
Patients with a diagnosis of major depressive disorder, who are currently either euthymic or mildly depressed, will be recruited for this study. 40 participants (ages 19-55) will be recruited from the community from two outpatient sites and 30 participants will be recruited from an inpatient site. For the outpatient sample, 20 patients will be recruited at University of British Columbia (UBC) and 20 patients will be recruited at Simon Fraser University (SFU), and for the inpatient sample, 30 patients will be recruited in collaboration with the John Volken Academy (JVA). Patients will complete an initial virtual assessment to assess eligibility, after which patients will complete the bWell cognitive assessment session. This session will include rating scales for current symptoms of depression/anxiety, subjective cognitive functioning, global/occupational functioning and a validated computerized neuropsychological test battery to assess objective cognitive functioning. Participants will complete a brief VR training session with the VR equipment. Subsequently, the bWell cognitive assessment program will be administered, followed by scales assessing tolerability and enjoyability/engagement.

Patients will then be randomized in a 1:1 ratio to receive bWell cognitive remediation or to a control group in which they passively experience various VR scenes. Randomization will occur separately in inpatient and outpatient groups. Patients are told that either method is hypothesized to have effects on their cognition and are therefore blinded to whether they are in the 'active' treatment group. Assessors for outcomes that are not self-reported or self-administered will also be blinded to group assignment. Participants randomized to the bWell cognitive remediation program will complete 40-minute remediation sessions using bWell twice a week for 8 weeks; the other group will view VR scenes in bWell without any instructed cognitive tasks. EEG recordings will be administered at baseline, at midpoint, and after completing the 8 weeks. At the end of the 8 weeks, measures of subjective cognitive functioning, global/occupational functioning and the computerized objective cognitive testing battery will also be repeated. Patients will also complete tolerability and enjoyment/engagement scales during the remediation procedure. Patients will be debriefed at the end of their participation about their treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* 19-55 years old
* Meeting the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for MDD as assessed by a standardized psychiatric interview (SCID-5-RV) conducted by a trained clinician.
* Patients will be euthymic or mildly depressed (defined by a Montgomery-Asberg Depression Rating Scale [MADRS] score < 19)
* Patients will report subjective cognitive deficits at baseline, as indicated by a total Perceived Deficits Questionnaire - Depression 20 [PDQ-D-20] score > 20 at study enrollment.
* If participants are on antidepressant therapy, participants will be on stable antidepressant therapy for at least 8 weeks prior to randomization. All concomitant doctor-prescribed medications must be at a stable dose for 4 weeks prior to the randomization visit.
* If participants are on psychotherapy, participants will be on stable adjunct psychotherapy for at least 12 weeks prior to randomization
* If comorbid diagnosis of attention deficit hyperactivity disorder (ADHD), patients must be on stable dose of stimulants for at least 8 weeks prior to randomization.
* Participants will be able to follow written and verbal instructions in English

Exclusion Criteria:

* Moderate - severely depressed patients will be excluded at this point due to acceptability concerns (e.g. potential for cybersickness)
* Presence of significant neurological disorders, head trauma, or other unstable medical conditions. These conditions may adversely impact cognitive functioning and influence study results.
* Presence of other psychiatric disorder (e.g. anxiety, psychotic disorder) that may be considered primary.
* Meeting DSM-5 criteria for alcohol or other substance use disorder within three months prior to the randomization visit.*
* Use of benzodiazepine medications more than three times per week and/or within 24 hours of baseline or close out visit
* Use of cannabis or alcohol within 24 hours, or tobacco within 30 minutes of baseline or close out visit

  * Patients recruited from the inpatient settings at the John Volken Academy, have a slightly different exclusion criteria for substance use disorders and only will be excluded if they meet DSM-5 criteria for alcohol or other substance use disorder within one month prior to the randomization visit.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | 8 weeks
  Measured separately in inpatient and outpatient settings, target of 2/month total from both sites. Will be assessed every 6 months and appropriate action taken if target not met.
Session completion rates | 8 weeks
  Measured separately in inpatient and outpatient settings, target of 80% completion of all studies. Will be assessed after the 5th and 10th participants to complete bWell-D assessment and mid-point of bWell-D remediation, with appropriate action taken if not met.
Study drop out rates | 8 weeks
  Measured separately in inpatient and outpatient settings, target 20% or less participant dropouts. Will be assessed after the 5th and 10th participants to complete bWell-D assessment and mid-point of bWell-D remediation, with appropriate action taken if not met.

SECONDARY OUTCOMES:
Change in cognitive functioning in active vs. control groups | 8 weeks
  Assessed using the Neurocognitive Index (NCI) score generated by the Central Nervous System Vital Signs (CNS-VS), an index of global cognitive functioning
Change in global psychosocial functioning in active vs. control groups | 8 weeks
  Assessed through self-report using the Sheehan Disability Scale (SDS) and Quality of Life Enjoyment and Satisfaction Questionnaire. When self-reporting scores on the SDS, patients are asked to rank on a 10-point scale the level of disruption they have experienced at work/school, in their social life and home responsibilities over the past week. Total scores range from a minimum of 0 to a maximum of 30, where higher scores represent increased functional impairment.
Change in individual cognitive domains in active vs. control groups | 8 weeks
  Assessed via the individual domain scores generated by the CNS-VS computerized battery
Change in subjective perceived cognitive functioning in active vs. control groups | 8 weeks
  Assessed via the Perceived Deficits Questionnaire for Depression (PDQ-D), a self-report scale assessing patients' perceived functioning in four domains: attention/concentration, planning/organization, retrospective memory and prospective memory. Total score ranges from 0 to 80, where higher scores represent increased cognitive impairment.
Measure of video game satisfaction/enjoyability of bWell-D remediation in active vs. control groups | 8 weeks
  Assessed using the The Game User Experience Satisfaction Scale-18 (GUESS-18). Total score ranges from a minimum value of 9 to a maximum value of 63, where higher scores represent increased satisfaction.
Change in occupational psychosocial functioning in active vs. control groups | 8 weeks
  Assessed through self-report using the Lam Employment Absence and Productivity Scale (LEAPS). When self-reporting on LEAPS, patients rate the degree to which problems with low energy/motivation, anxiety/irritability, poor concentration, decreased productivity/mistakes and interpersonal problems have impacted their occupational performance over the past 2 weeks. Total scores range from a minimum of 0 to a maximum of 28, where higher total scores represent increasingly impaired professional functioning.
Change in subjective everyday cognitive functioning in active vs. control groups | 8 weeks
  Assessed via the Cognitive Failures Questionnaire (CFQ), which assesses lapses of attention, perception and memory in real-life. Total score ranges from a minimum of 0 to a maximum of 100, where higher scores represent increased everyday cognitive failures.
Measure of engagement with bWell-D remediation in active vs. control groups | 8 weeks
  Assessed using the User Engagement Scale (UES). There is a minimum score of 0 and a maximum score of 235.62, where higher scores represent increased engagement.
Measure of tolerability of bWell-D remediation in active vs. control groups | 8 weeks
  Assessed using Simulator Sickness Questionnaire (SSQ). Patients rate the presence and severity of various symptoms of cybersickness, including nausea and ocular discomfort. There is a minimum score of 4 and a maximum score of 20, where higher scores represent increased simulator sickness.

CONTACTS AND LOCATIONS:
Overall Officials: Trisha Chakrabarty, MD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gagnon Shaigetz V, Proulx C, Cabral A, Choudhury N, Hewko M, Kohlenberg E, Segado M, Smith MSD, Debergue P. An Immersive and Interactive Platform for Cognitive Assessment and Rehabilitation (bWell): Design and Iterative Development Process. JMIR Rehabil Assist Technol. 2021 Nov 3;8(4):e26629. doi: 10.2196/26629. PMID 34730536
- [Background] Hernandez Hernandez ME, Michalak E, Choudhury N, Hewko M, Torres I, Menon M, Lam RW, Chakrabarty T. Co-design of a Virtual Reality Cognitive Remediation Program for Depression (bWell-D) With Patient End Users and Clinicians: Qualitative Interview Study Among Patients and Clinicians. JMIR Serious Games. 2023 Apr 7;11:e43904. doi: 10.2196/43904. PMID 37027183